CLINICAL TRIAL: NCT07403903
Title: Having an Amazing Start? A Randomized Controlled Trial Evaluating the Effectiveness of a Parenting Intervention
Brief Title: Amazing Start Parenting Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chow Tai Fook Charity Foundation (Unknown); Lee Hysan Foundation (Unknown)
Responsible Party: Principal Investigator, Wong Tin Yau, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EA230380
Record Dates: First submitted 2026-02-04; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Parenting Intervention
Keywords: Child development; Parenting; Well-being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Amazing start parenting intervention
  Interventions: Behavioral: Amazing start parenting intervention
- Control (No Intervention): • No service is provided to the families in the control group

INTERVENTIONS:
Behavioral: Amazing start parenting intervention — * 14 session on Parent-child Play Group
  * 14 session on 1 on 1 Playdate cum Parent-child Play-based Coaching
  * 6 session on Mentorship & Parents Social Network
  * 4-6 session on Parents' Wellness Program
  * 2 Amazing Start Boxes
  Arms: Intervention

SUMMARY:
Whether young children can develop healthily depends a lot on the family environment where they grow up in. Risk factors, such as low family income or health issues within the family, may pose threats to young children's development. To mitigate the effects of these risk factors, the research team has developed a community parenting program titled "Amazing Start", which aims to improve young children's well-being through the provision of parenting interventions to the families with known risk factors. The parenting interventions include one-to-one coaching on parent-child interactions as well as parent support groups that are led by social workers. This 2-year study aims to investigate the effectiveness and sustainability of the "Amazing Start" community parenting intervention program for at-risk families across three districts in Hong Kong using a randomized controlled trial. Participating families are randomized to either the experimental group, where parenting interventions are provided for a period of 9 months, or the wait-list control group, where no parenting intervention is provided during this 9-month period. Pre-test and post-test are conducted to assess the development of young children, as well as the parental stress, parental sense of competence, and parental satisfaction of the participating families. The wait-list control group receives the parenting intervention after the post-test.

DETAILED DESCRIPTION:
There are strong relations between children's family background and their development. Infants and toddlers growing up in single-parent families, low-income families, and families with members having physical or mental health issues are less likely to meet developmental milestones at appropriate times compared to their peers who grow up in intact, well-off, and healthy families. The lack of parenting knowledge and skills is one of the potential factors that may explain the relation between children's family background and their development. Infants and toddlers growing up in at-risk families may face more stressors, and they may not have the means to acquire relevant parenting knowledge and skills that are important for children's development. Intervention programs that target parenting skills may help mitigate the negative effects of these risk factors on children's development.

Observing this service gap, the research team has developed a parenting program titled "Amazing Start". The program aims to improve infants' and toddlers' development through improving parents' parenting skills and reducing their parental stress. These interventions involve one-to-one coaching on parent-child interactions as well as parent support groups that are led by social workers. The intervention is delivered to those who have 2 or more of the risk factors listed below: (1) single-parent family, (2) ethnic minority, (3) new parents, (4) low-income family, (5) families with newborn twins, (6) persistent family conflicts, and (7) family members suffering from long-term illness.

A randomized controlled trial will be conducted to examine the effectiveness of the intervention. Families who are identified as having at least 2 risk factors will be randomly assigned to one of the two conditions. Families assigned to the experimental condition will receive the intervention for nine months, while families assigned to the wait-list control condition will not receive any services during this period. Pre-test and post-test will be conducted to assess the program's effectiveness in improving parental sense of competence, reducing parental stress, enhancing parents' satisfaction about parenting, as well as promoting infants' and toddlers' development. The wait-list control group will receive the parenting intervention after the post-test.

ELIGIBILITY:
Inclusion Criteria:

* 1. Families with infants and toddlers aged 0 to 36 months
* 2. Families residing in Kwun Tong, Yuen Long, and Yau Tsim Mong Districts
* 3. Families with at least 2 risk factors listed below

  1. single-parent family,
  2. ethnic minority,
  3. new parents,
  4. low-income family,
  5. families with newborn twins,
  6. persistent family conflicts, and
  7. family members suffering from long-term illness

Exclusion Criteria:

* Families with fewer than 2 risk factors listed above

Ages: 0 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 270 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Child development | 9 months after the start of the intervention
  Ages and stages questionnaire - third edition (ASQ-3). The ASQ-3 is a brief screening tool for assessing young children's (aged 1 to 66 months) development in five different domains, namely communication, gross motor, fine motor, problem solving, and personal-social. There are 6 items in each domain. Each item involves a simple task in which the child needs to complete with the relevant materials. As the ASQ-3 consists of different items for children of different age, the number of domains reaching the appropriate developmental milestones will be used as an overall indicator of the child's development.

SECONDARY OUTCOMES:
Parenting sense of competence | 9 months after the start of the intervention
  Parenting sense of competence scale (Gibaud-Wallston & Wandersman, 1978; Ngai, et al., 2007). This is a 17-item 6-point Likert scale assessing parents' sense of competence. Total score is used in the analysis.
Parental stress | 9 months after the start of the intervention
  Parental stress scale (Berry and Jones, 1995; translated to Chinese by Cheung, 2000). This is a 17-item 6-point Likert scale assessing parental stress. Total score is used in the analysis.
Parents' life satisfaction | 9 months after the start of the intervention
  Satisfaction level on different life aspects. This is a self-report life satisfaction questionnaire developed by the research team. It covers various aspects ranging from parent's attitude towards parent-child interactions, the mastery of parenting knowledge and skills, family interaction patterns, as well as self-control of emotions. Each domain is rated along a 11 point Likert scale, ranging from 0 (very unsatisfactory) to 10 (very satisfactory). Total score is used in the analysis.
Cost effectiveness | 48 months after the start of the intervention
  After the intervention, the research team will obtain information about the cost of service delivery in order to calculate the cost-effectiveness of the program. Cost-effectiveness of the parenting program versus control will be assessed and expressed in terms of incremental cost per one unit gain in effectiveness.

CONTACTS AND LOCATIONS:
Locations (1):
- The Univesity of Hong Kong, Hong Kong, Region, Hong Kong

IPD SHARING:
Plan to Share IPD: No